CLINICAL TRIAL: NCT06066866
Title: Microbiome Sampling in GI Disease With a Focus on Small Intestinal Microbial Assessment
Status: Not yet recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Spencer, Instructor, Stanford Gastroenterology and Hepatology, Stanford University
Other Study IDs: 71429
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Healthy; IBS - Irritable Bowel Syndrome; Inflammatory Bowel Diseases
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: endoscopic sampling of luminal fluid — We will collect luminal fluid via endoscopic sampling

SUMMARY:
GI disorders are influenced by the gut microbiome. To date, sampling of the small intestine in GI disorders has been limited. The investigators plan to sample the small intestinal contents during endoscopy for research purposes.

DETAILED DESCRIPTION:
Current guidelines (AGA Clinical Practice Update, 2020) report the definition of SIBO as a clinical entity lacks precision and consistency; it is a term generally applied to a clinical disorder where symptoms, clinical signs, and/or laboratory abnormalities are attributed to changes in the numbers of bacteria or in the composition of the bacterial population in the small intestine. To date, there is unlimited knowledge regarding the diagnostic criterion which has been limited by nonspecific and nonsensitive testing such as breath tests. Breath tests have a limited use in patients with IBS-D who inherently have increased gut transit time rendering the testing invalid for accurately measuring small intestinal bacteria. Additionally, the relationship between SIBO and symptoms in patients without obvious risk factors (such as anatomical changes due to surgery) is unknown. The investigators study aims to investigate the microbial landscape of the small intestine in healthy patients and those with GI disease (suspected or diagnosed) undergoing an upper endoscopy by collecting an aspirate of patient small intestinal fluid and studying it.

ELIGIBILITY:
Inclusion Criteria:

* Age >18years
* Patients seen at Stanford University Digestive Health Center who are scheduled for an upper endoscopy as part of their Standard Of Care

Exclusion Criteria:

Children (under age 18years) Pregnant Women and Fetuses Neonates (0 - 28 days) Impaired Decision Making Capacity

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen at Stanford University Digestive Health Center who are scheduled for an upper endoscopy as part of their Standard Of Care
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Ability to isolate live bacteria from 95% of samples | 1-4 years
  We aim to isolate live bacteria from 95% of samples

SECONDARY OUTCOMES:
Ability to measure quantitative Colony Forming Units (CFUs) in 90% of samples | 1-4 years
  We aim to measure quantitative Colony Forming Units (CFUs) in 90% of samples

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Spencer, MD,PhD, Principal Investigator — Stanford University; Linda A Nguyen, MD, Study Chair — Stanford University

IPD SHARING:
Plan to Share IPD: No